CLINICAL TRIAL: NCT05960474
Title: Coronary Microvascular Disease (CMD) Registry
Status: Recruiting | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CMDR
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Coronary Microvascular Dysfunction
MeSH Terms: interventions — Treatment Outcome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Outcomes for Patients with CMD — Our objective is to perform a retrospective/prospective descriptive study on the short term to longterm (up to 5 years of follow-up) outcomes of patients with coronary microvascular disease diagnosis invasively

SUMMARY:
The purpose of this project is to provide appropriate administrative and technical supports for the warehousing and use of a database of patients with coronary microvascular disease (CMD). This protocol will outline the process for identification and capture of data, storage, as well as data use and sharing internally and externally for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Those with Coronary Microvascular Disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects to be enrolled in either objective for this registry includes patients, 18 years or older, with coronary microvascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Establish a Registry of CMD patients | 10 years

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Memorial Regional Hospital, Hollywood, Florida
  - MedStar Southern Maryland, Clinton, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Qaraghuli A, Chitturi KR, Kumar S, Cellamare M, Ozturk S, Sawant V, Zhang C, Verma BR, Galo J, Chaturvedi A, Ben-Dor I, Satler L, Rogers T, Waksman R, Hashim H, Case BC. Exploring the impact of age on microvascular function: Insights from the Coronary Microvascular Disease Registry. Int J Cardiol. 2026 Jan 1;442:133858. doi: 10.1016/j.ijcard.2025.133858. Epub 2025 Sep 2. PMID 40907829
- [Derived] Abusnina W, Merdler I, Cellamare M, Chitturi KR, Chaturvedi A, Feuerstein IM, Zhang C, Ozturk ST, Deksissa T, Sawant V, Lopez K, Lupu L, Haberman D, Ben-Dor I, Satler LF, Waksman R, Hashim HD, Case BC. Epicardial Fat Tissue: A Potential Marker for Coronary Microvascular Dysfunction. J Am Heart Assoc. 2025 Feb 4;14(3):e038484. doi: 10.1161/JAHA.124.038484. Epub 2025 Feb 3. PMID 39895522
- [Derived] Chitturi KR, Kumar S, Frisancho FT, Rahman S, Verma BR, Cellamare M, Merdler I, Ozturk ST, Cermak V, Sawant V, Zhang C, Ben-Dor I, Waksman R, Hashim HD, Case BC. The Prevalence of Coronary Microvascular Dysfunction in Patients With Type 2 Diabetes Mellitus. Catheter Cardiovasc Interv. 2025 Apr;105(5):1120-1123. doi: 10.1002/ccd.31429. Epub 2025 Jan 29. PMID 39888248
- [Derived] Chitturi KR, Kumar S, Hill AP, Lorente-Ros M, Cellamare M, Merdler I, Abusnina W, Haberman D, Lupu L, Chaturvedi A, Ozturk ST, Cermak V, Sawant V, Zhang C, Ben-Dor I, Tsimploulis A, Waksman R, Hashim HD, Case BC. Prevalence of Arrhythmias in Patients With Coronary Microvascular Dysfunction. Catheter Cardiovasc Interv. 2025 Feb;105(2):483-490. doi: 10.1002/ccd.31324. Epub 2024 Dec 11. PMID 39660783
- [Derived] Merdler I, Bazarbashi N, Medranda GA, Zhang C, Ozturk ST, Sawant V, Ben-Dor I, Waksman R, Hashim HD, Case BC. Comparing planned versus ad hoc coronary microvascular assessment: Early findings from the Coronary Microvascular Disease Registry. Cardiovasc Revasc Med. 2024 Oct;67:69-74. doi: 10.1016/j.carrev.2024.04.017. Epub 2024 Apr 12. PMID 38724408
- [Derived] Case BC, Merdler I, Medranda GA, Zhang C, Ozturk ST, Sawant V, Garcia-Garcia HM, Satler LF, Ben-Dor I, Hashim HD, Waksman R. Coronary Microvascular Disease Registry (CMDR): Study design and rationale. Cardiovasc Revasc Med. 2024 Sep;66:63-67. doi: 10.1016/j.carrev.2024.03.021. Epub 2024 Mar 27. PMID 38631936
- [Derived] Merdler I, Wallace R, Banerjee A, Medranda GA, Reddy P, Cellamare M, Zhang C, Ozturk ST, Sawant V, Lopez K, Ben-Dor I, Waksman R, Case BC, Hashim HD. Coronary microvascular dysfunction assessment: A comparative analysis of procedural aspects. Catheter Cardiovasc Interv. 2024 Apr;103(5):703-709. doi: 10.1002/ccd.30990. Epub 2024 Mar 23. PMID 38520176